CLINICAL TRIAL: NCT02241265
Title: Spirometric Response to Bronchial Thermoplasty in Patients With Severe Asthma
Status: Recruiting | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 3790; 3790 (Other: OUHSC IRB)
Record Dates: First submitted 2014-05-05; First posted 2014-09-16 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Asthma
Keywords: asthma; thermoplasty
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Past Bronchial Thermoplasty data: Data will be collected from records of patients who, in the past, have undergone bronchial thermoplasty.

SUMMARY:
The investigators hypothesis is that there will be improvement in FEV1 in patients with severe asthma. This is a retrospective data study that reviews preexisting medical records; no patients will be enrolled.

DETAILED DESCRIPTION:
The investigators plan is to retrospectively evaluate spirometry on patients with severe asthma who have undergone bronchial thermoplasty. The procedure will have been done according to the recommended protocol of three separate sessions. For each patient all available spirometric data obtained before and after thermoplasty will be used. Data will be collected from two centers, OU Medical Center and St. Francis Hospital in Tulsa, OK. All procedures done at St. Francis have been performed by a single physician and he is providing their spirometric data for the investigators study. The following data will be collected for all participants undergoing bronchial thermoplasty: Age, height, sex, weight, medical history, smoking history, baseline spirometry before and after bronchodilators, post thermoplasty spirometry before and after bronchodilators.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* severe asthma diagnosis
* decreased FEV1

Exclusion Criteria:

* < 18 years of age

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective review of Asthma Patients' records
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The primary endpoints are improvements in prebronchodilator FEV1 and FVC. | 1 year after thermoplasty
  The primary endpoints are improvements in prebronchodilator FEV1 and FVC by 12% predicted.

SECONDARY OUTCOMES:
Secondary endpoints are improvements in postbronchodilator FEV1 and FVC and degree of bronchodilator responsiveness. | 1 year after thermoplasty
  Secondary endpoints are improvements in postbronchodilator FEV1 and FVC and degree of bronchodilator responsiveness by 12% predicted.

CONTACTS AND LOCATIONS:
Overall Officials: Brent Brown, MD, Principal Investigator — OUHSC
Locations (1):
- OUHSC, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data may only be shared upon review of OUHSC Legal office and IRB. Data sharing agreement required. Contact research@ouhsc.edu to initiate data requests. No personally identifiable data will be shared.